CLINICAL TRIAL: NCT06067880
Title: Surgical Intervention and Post Operative Improvement in Patients With Lymphatic Diseases.
Brief Title: Surgical Intervention and Lymphatic Diseases.
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202201453B0
Record Dates: First submitted 2023-09-28; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lower Limb Lymphedema: This was a retrospective cohort propensity score-matched study. Patients with cancer-related unilateral lower limb lymphedema were enrolled.
  Interventions: Other: Cancer-related Unilateral; Other: Normal + Ectasis LVs

INTERVENTIONS:
Other: Cancer-related Unilateral — This group included patients who have used only contraction type LVs.
Other: Normal + Ectasis LVs — This group included patients who had only non- contraction type LVs.

SUMMARY:
Supermicrosurgical LVA has been proven effective in treating moderate to severe lymphedema, including cases with diffuse dermal backflow (DB) and even severe lymphatic fluid leakage. Therefore, the use of LVA should not be limited to mild lymphedema, and its indications should be expanded to become a primary surgical approach for more severe lymphedema cases. Among all surgical procedures for lymphedema, LVA is the least invasive, allowing for rapid recovery, minimizing the complications, and reducing medical costs.

DETAILED DESCRIPTION:
Lymphatic-related diseases such as lymphedema often result from damage to the lymphatic system due to tumor removal and lymph node dissection surgeries, as well as tissue fibrosis caused by post-operative radiation therapy. This can lead to obstruction in the proximal channels of lymphatic flow, resulting in swelling, deformity of the distal limbs, poor wound healing, or cellulitis.

In the case of lymphatic-related diseases like lymphedema, improvement can be achieved through surgical interventions. Surgery can be categorized into physiologic reconstruction and volume reduction procedures. Among them, Supermicrosurgical Lymphaticovenous Anastomosis (LVA) is a form of physiologic reconstruction. LVA involves the separation of lymphatic vessels in the affected limb and their anastomosis with nearby small veins to alleviate limb swelling and reduce the risk of cellulitis. When using lymphaticovenous bypass surgery to treat lymphedema, the ideal scenario is to use veins for anastomosis that do not have venous blood reflux. This is because veins generally have higher blood pressure than lymphatic fluid, and if venous blood flows into the lymphatic vessels over the long term, it can reduce the patency of the lymphaticovenous anastomosis site. The choice of anastomosis technique, based on the size and position of the lymphatic vessels and veins, can also impact the post-operative outcomes. Therefore, factors such as lymphatic vessel size, flow rate, function, vein size, pressure, and the presence of reflux are closely related to the success of lymphaticovenous bypass surgery.

Supermicrosurgical LVA has been proven effective in treating moderate to severe lymphedema, including cases with diffuse dermal backflow (DB) and even severe lymphatic fluid leakage. Therefore, the use of LVA should not be limited to mild lymphedema, and its indications should be expanded to become a primary surgical approach for more severe lymphedema cases. Among all surgical procedures for lymphedema, LVA is the least invasive, allowing for rapid recovery, minimizing the complications, and reducing medical costs.

ELIGIBILITY:
Inclusion Criteria:

* This study including patients diagnosed with lymphatic-related diseases at Kaohsiung Chang Gung Memorial Hospital from September 1, 2015, to August 31, 2022.

Exclusion Criteria:

* Patients under the age of 20.
* Patients with incomplete medical records.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients (age >20 years) receiving LVA for gynecologic cancer-related unilateral lower limb lymphedema at a tertiary medical center were retrospectively reviewed from October 2015 to July 2022.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2022-09-23 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Volume change after LVA. | 6/12 months
  The primary endpoint was the volume change at 6/12 months after LVA.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Derived] Knoz M, Wang YM, Luo SD, Wu SC, Lin WC, Tsai PY, Chien PC, Hsieh CH, Yang JC. Comparison of contraction-type and noncontraction-type lymphatic vessels in lymphaticovenous anastomosis for cancer-related unilateral lower limb lymphedema: a retrospective cohort propensity-score-matched outcome analysis. Int J Surg. 2024 Apr 1;110(4):1913-1918. doi: 10.1097/JS9.0000000000001106. PMID 38265436